CLINICAL TRIAL: NCT01111266
Title: Evaluation of Performance and Safety Profile of Xevonta High Flux Dialyzer With Special Focus on Determination of in Vivo Ultrafiltration Coefficient in Patients With CKD
Brief Title: Determination of in Vivo Ultrafiltration Coefficient (KUF) in Patients With Chronic Kidney Disease (CKD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.Braun Avitum AG (Industry)
Collaborators: Labor Limbach, Heidelberg, Germany (Unknown); Clin-Sol, Würzburg, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BA-I-H-09-02
Record Dates: First submitted 2010-04-15; First posted 2010-04-27 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Kidney Disease
Keywords: in vivo KUF; ß2M; leptin
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: xevonta — Patients will be treated with 3 different sizes of xevonta (2 weeks each size) for determination of in vivo KUF following "FDA Guidance for the Content of Premarket Notifications for Conventional and High Permeability Hemodialyzers". In addition blood samples will be collected for determination of removal rates of different small molecules and protein.

SUMMARY:
The purpose of this study is to determine the in-vivo ultrafiltration coefficient for different sizes of xevonta High-Flux dialyzers following FDA guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from patient or parents/ guardian.
* Subject age >= 18
* Effective blood flow 350 ml/min and dialysate flow of 500 ml/min
* On hemodialysis for a minimum of 3 months
* Use of Cimino- or Gore-tex shunts
* Routine dialysis-treatment for 240 min
* Documented dialysis adequacy parameter that has been stable for past 3 months
* Plan to dialyze at participating hemodialysis centre for at least 3-months duration.
* Free from any currently known unusual clotting or access problems
* Hepatitis B surface antigen (HbsAg) negative, documented within the past 90 days or Hepatitis B surface antibody (anti-HBs) positive.
* Anti Hepatitis C Virus (Anti-HCV) negative, documented within the past 90 days
* Anti Human Immunodeficiency Virus (Anti HIV) negative, documented within the past 90 days
* Hematocrit (HCT) between 25 and 40% or haemoglobin (Hb) not less than 8 g/dL, as documented 14 days prior to the first treatment

Exclusion Criteria:

* Patients who are unable to tolerate an effective blood flow of 350 ml/min
* Patients using catheter for dialysis
* Pregnant or nursing woman. Women of childbearing potential must agree to avoid pregnancy during the study period by use of hormonal contraception (implantable; patch; oral) and/ or double-barrier methods (any double combination of: IUD; condom with spermicidal gel; diaphragm; sponge; cervical cap)
* Previous plan for extended absences from the participating hemodialysis centre
* Expected to be transplanted (living related donor) within the maximum of 3 months for the study period
* Any serious medical conditions or disability, which in the opinion of the investigator, would interfere with treatment or assessment or preclude completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
in vivo KUF | 6 weeks
  The objective of this study is to to determine in vivo KUF for three different sizes (1.2; 1.8 and 2.3 m^2) of xevonta High-Flux to compare obtained data with respective in vitro KUF data.

SECONDARY OUTCOMES:
Determination of removal rates | 6 weeks
  Removal rates for urea, phosphate, creatinine, albumin, leptin and Beta2-microglobulin will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Wagner, Prof. Dr., Study Director — B.Braun Avitum AG
Locations (1):
- Georg-Haas Dialysezentrum der PHV, Giessen, Hesse, Germany